CLINICAL TRIAL: NCT00920062
Title: Ultrasound Dilution Measurement of Recirculation During Venovenous Extracorporeal Membrane Oxygenation
Brief Title: Measurement of Recirculation During Venovenous Extracorporeal Membrane Oxygenation (VV ECMO)
Status: Completed | Type: Observational
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: TSI-C-HCE101-3A-H; 2R44HL082022-02 (NIH)
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Venovenous Extracorporeal Membrane Oxygenation; Recirculation
Keywords: recirculation; ultrasound dilution; venovenous extracorporeal membrane oxygenation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to test the usefulness of ultrasound dilution recirculation measurements in patients receiving venovenous extracorporeal membrane oxygenation as therapy. The ultrasound dilution measurements determine the efficiency of support provided by venovenous extracorporeal membrane oxygenation. At the present time there are no other devices available to make recirculation measurements.

DETAILED DESCRIPTION:
At the present time there are no devices available to measure recirculation in patients on venovenous extracorporeal membrane oxygenation. The study uses an external monitor, laptop computer, clamp on flowsensors and ultrasound dilution technology to measure blood flow. Measurements are made by injecting 0.5 - 1 ml/kg of sterile isotonic saline into the patient's extracorporeal circuit. The subject will be monitored throughout the measurements. The measurements will be coordinated with the regular care of the patient and their extracorporeal circuit.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 0 and 21 years of age
* Patients receiving venovenous extracorporeal membrane oxygenation as treatment.

Exclusion Criteria:

* Patients over 21 years of age
* Patients not receiving venovenous extracorporeal membrane oxygenation.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Neonatal and/or pediatric patients receiving venovenous extracorporeal membrane oxygenation as treatment.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2007-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Recirculation measurements made in patients receiving venovenous extracorporeal membrane oxygenation. | Duration of venovenous extracorporeal membrane oxygenation

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai M Krivitski, PhD, DSc, Principal Investigator — Transonic Systems Inc.; Bonnie L Marr, MD, Principal Investigator — Crouse Hospital
Locations (1):
- Crouse Hospital, Syracuse, New York, United States

REFERENCES:
- [Background] Clements D, Primmer J, Ryman P, Marr B, Searles B, Darling E. Measurements of recirculation during neonatal veno-venous extracorporeal membrane oxygenation: clinical application of the ultrasound dilution technique. J Extra Corpor Technol. 2008 Sep;40(3):184-7. PMID 18853830